CLINICAL TRIAL: NCT00123890
Title: A Screening Protocol to Determine Eligibility for One of Three Phase III Treatment Studies Evaluating the Efficacy and Safety of GW873140 in R5-tropic and R5/X4-tropic HIV-1 Infected, Treatment-experienced Subjects With Drug-resistant Virus or an Observational Study.
Brief Title: Screening Protocol To Determine Eligibility For Studies Of The Chemokine Coreceptor 5 (CCR5) Antagonist GW873140
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to hepatoxicity of compound
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Masking: None | Purpose: Diagnostic
Other Study IDs: CCR104627
Record Dates: First submitted 2005-07-22; First posted 2005-07-26 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: HIV Infection
Keywords: HIV-1 GW873140 CCR5 antagonist experienced
MeSH Terms: conditions — HIV Infections | interventions — aplaviroc

INTERVENTIONS:
Drug: GW873140

SUMMARY:
The purpose of this study is to determine eligibility for one of three treatment studies of the CCR5 antagonist GW873140 or an observational study without GW873140. No investigational treatment will be administered through this study.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected.
* Screening viral load at least 5000copies/mL.
* Total prior antiretroviral experience of at least 3 months and documented resistance to at least one drug in each of the following classes: nucleoside reverse transcriptase inhibitors (NRTI), non-nucleoside reverse transcriptase inhibitors (NNRTI), and protease inhibitors (PI), stable antiretroviral regimen (or no antiretroviral treatment) for at least 4 weeks before screening.
* Able to receive a ritonavir-boosted protease inhibitor during treatment studies.
* Women of childbearing potential must use specific forms of contraception.

Exclusion criteria:

* Acute laboratory abnormalities.
* History of pancreatitis or hepatitis, hepatitis B or hepatitis C coinfection, or any chronic liver disease. Screening liver function tests will be used to determine eligibility.
* Changes to antiretroviral therapy from 4 weeks prior to screening until Day 1 of treatment or observational studies.
* Pregnancy or breastfeeding women.
* Recent participation in an experimental drug trial.
* Prior use of a CCR5 or CXCR4 antagonist.
* Significant ECG abnormalities or significant history of active pancreatitis, hepatitis, opportunistic infections, malabsorption disorders, cancer, or severe illness.
* Current use of certain medications may exclude participation in this study.
* Additional qualifying criteria and laboratory test requirements to be assessed by study physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-06; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Determination of subject eligibility for CCR102709, CCR104456, CCR104458, or CCR104629.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Ph.D., Study Director — GlaxoSmithKline
Locations (41):
- United States (33):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Laguna Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Tarzana, California
  - GSK Investigational Site, Glastonbury, Connecticut
  - GSK Investigational Site, Norwalk, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Oakland Park, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, East Orange, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Hampton, Virginia
  - GSK Investigational Site, Lynchburg, Virginia
  - GSK Investigational Site, Spokane, Washington
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Charleroi
- GSK Investigational Site, Toronto, Ontario, Canada
- GSK Investigational Site, Copenhagen, Denmark
- Germany (4):
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia